CLINICAL TRIAL: NCT04371640
Title: A Randomized, Double-Blinded, Placebo-Controlled Trial Evaluating the Virological Efficacy, Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Sirolimus Adjuvant Therapy in Patients With Coronavirus Disease (COVID-19)
Brief Title: Sirolimus in COVID-19 Phase 1
Acronym: SirCO-1
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Study population not regularly admitted to hospital and approaches have shifted away from repurposing old drugs.
Sponsor: Walter K. Kraft (Other)
Responsible Party: Sponsor-Investigator, Walter K. Kraft, Principal Investigator, Thomas Jefferson University
Organization: Thomas Jefferson University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 15680
Record Dates: First submitted 2020-04-28; First posted 2020-05-01 (Actual); Last update posted 2021-12-03 (Actual); Status verified 2021-12

CONDITIONS: SARS-CoV-2; Covid-19
MeSH Terms: conditions — COVID-19 | interventions — Sirolimus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Sirolimus (Active Comparator): Sirolimus + standard medical care Day 1: 10mg Days 2-7: 5mg
  Interventions: Drug: Sirolimus 1 MG/ML
- Placebo (Placebo Comparator): Placebo + standard medical care Day 1: 10mL Days 2-7: 5mL
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sirolimus 1 MG/ML — Oral solution
  Other Names: Rapamune
  Arms: Sirolimus
Drug: Placebo — Oral solution
  Arms: Placebo

SUMMARY:
This is a double-blinded, two-arm, randomized, placebo controlled study comparing the virological efficacy of add-on sirolimus with standard care to placebo and standard care. Virological efficacy is defined as the change from baseline to day 7 in SARS-CoV-2 viral burden measured by quantitative real-time polymerase chain reaction.

ELIGIBILITY:
Inclusion Criteria:

* Male or non-pregnant female >/=18 and </=65 years of age at the time of consent
* Laboratory confirmed SARS-CoV-2 infection
* Investigator-estimated hospitalization duration of at least 5 days

Exclusion Criteria:

* Need for >4 liters nasal cannula oxygen to maintain oxygen saturation >90%
* Hypersensitivity to sirolimus
* Pregnant or breastfeeding
* Anticipated transfer to another study hospital within 72 hours
* Alanine transaminase (ALT) >3 times the upper limit of normal
* Creatinine clearance <30mL/min as estimated by Cockcroft-Gault
* Underlying immunosuppression due to daily >5 mg prednisone equivalent a day, prior solid organ transplant, or other immunosuppression deemed by investigator to be potentially unsafe
* Co-administration with strong inhibitors of CYP3A4 and/or P-glycoprotein (P-gp) (such as ketoconazole, voriconazole, itraconazole, telithromycin, clarithromycin and others)
* Co-administration with strong inducers of CYP3A4 and/or P-glycoprotein (P-gp) (such as phenytoin or rifampin)
* Anticipated surgery within 1 month
* Need for healing of a fracture or a significant soft tissue wound

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-07-06 (Actual); Primary Completion 2021-07-30 (Actual); Study Completion 2021-07-30 (Actual)

PRIMARY OUTCOMES:
Change in SARS-CoV-2 viral burden from baseline to day 7 of treatment | Baseline, and days 1, 2, 3, 4, 5, 6, & 7 post-dose for all patients
  SARS-CoV-2 viral burden will be quantified for both arms using a qRT-PCR

SECONDARY OUTCOMES:
Change in SARS-CoV-2 viral burden at days 1-6 | Days 1, 2, 3, 4, 5, and 6 post-dose for all patients
  SARS-CoV-2 viral burden will be quantified for both arms using a qRT-PCR
Rate of treatment emergent adverse events | Days 1, 2, 3, 4, 5, and 6 post-dose for all patients
  Safety and tolerability of sirolimus in patients with COVID-19

CONTACTS AND LOCATIONS:
Overall Officials: Walter K Kraft, MD, Principal Investigator — Thomas Jefferson University
Locations (1):
- Thomas Jefferson University Hospital, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No